CLINICAL TRIAL: NCT06098794
Title: The Effects of Sodium Bicarbonate Supplementation on Intense Exercise Performance
Brief Title: Effect of Sodium Bicarbonate on Exercise Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Motricidade Humana (Other)
Responsible Party: Principal Investigator, Cristina Monteiro, Assistant Professor, Faculdade de Motricidade Humana
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: RepSprintsSodiumBicarbonate
Record Dates: First submitted 2023-10-06; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Sodium Bicarbonate
Keywords: Ergogenic Dietary Supplement; Repeated Sprints Performance; Muscle Oxygenation; Oxygen Consumption
MeSH Terms: interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Bicarbonate - Placebo (Experimental): First exercise performance assessment after ingesting sodium bicarbonate. Second exercise performance assessment after ingesting placebo
  Interventions: Dietary Supplement: Sodium Bicarbonate; Dietary Supplement: Placebo
- Placebo - Sodium Bicarbonate (Experimental): First exercise performance assessment after ingesting placebo. Second exercise performance assessment after ingesting sodium bicarbonate
  Interventions: Dietary Supplement: Sodium Bicarbonate; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Sodium Bicarbonate — Capsules containing 0.3 g/kg of body weight of sodium bicarbonate were ingested in two doses. The first intake (0.2 g/kg) was performed together with a carbohydrate-enriched meal 2 h before a repeated sprint exercise protocol, and the second (0.1 g/kg) occurred 1 h later.
Dietary Supplement: Placebo — Capsules containing 0.3 g/kg of body weight of celulose were ingested in two doses. The first intake (0.2 g/kg) was performed together with a carbohydrate-enriched meal 2 h before a repeated sprint exercise protocol, and the second (0.1 g/kg) occurred 1 h later.

SUMMARY:
This was a randomized, double-blind, placebo controlled, crossover trial. The study aimed to assess the effect of sodium bicarbonate on the ability to perform a repeated sprint task by female football players. The researches hypothesis was that sodium bicarbonate increases the ability to remove lactic acid from muscle cells reducing its intracellular accumulation and increasing energetic efficiency resulting in the increase of peak power output, mean power output, or total work or in the decrease of the sprint decrement in each set of the repeated sprints task.

DETAILED DESCRIPTION:
Experimental design: The study consisted of a randomized, double-blind, controlled, crossover trial where 11 female football players performed, in a randomized order, two repeated sprints tasks in a cycle ergometer, after having ingested either sodium bicarbonate (SB) or placebo (PL). Body composition of the athletes was characterized by bioelectrical impedance analysis with a single frequency (50 kHz) device (BIA 101 Anniversary, Akern, Florence, Italy) before the exercise sessions. Data collection was separated by a period of at least one week within a period of time not exceeding one month and performed at the same time of the day for each participant. Data regarding performance, blood lactate accumulation, pulmonary gas exchange, heart rate (HR), muscle oxygenation and neuromuscular fatigue were collected during these two sessions.

Supplementation protocol: The participants ingested capsules containing 0.3 g/kg of body weight of SB or cellulose as PL divided into two doses. The first intake (0.2 g/kg) occurred 2 h before the beginning of the protocol, and the second (0.1 g/kg) occurred 1 h later. Possible gastrointestinal symptoms associated with supplement ingestion were controlled with a questionnaire based on the questionnaire applied by Miller et al. (2016).

Repeated sprints protocol: The RSA protocol was performed in a cycle ergometer (Monark Ergomedic 894 E, Monark Exercise AB, Vansbro, Sweden) and was composed of 3 sets of 6 sprints with 6 s duration with a workload of 4% of the body mass. Repetitions were separated by 24 s of active recovery, and participants were conceded 5 min of passive recovery to rest between sets. The protocol was preceded by a 5-min warm-up in which athletes pedalled at a speed of 60 to 70 rpm.

Performance Measurements: Performance was evaluated by monitoring peak power output, mean power output, total work and the sprint decrement in each set of the two repeated sprints task.

Blood lactate accumulation: Lactate concentration was assessed (Lactate Pro 2, KDK Corporation, Kyoto, Japan) in capillary blood from the ear lobe before the beginning of each protocol, 1 min after the end of each set, and at min 1 and every 2 min after the tasks were completed, until the value started to decrease. At the end of the tasks, the maximal values achieved were considered for analysis.

Pulmonary gas exchange and heart rate: Oxygen uptake, carbon dioxide production and ventilation (VO2, VCO2, VE, respectively) were measured breath-by-breath, during the protocol, using a gas analyser (MetaMax 3B, Cortex Biophysik, Leipzig, Germany). Heart rate was continuously evaluated using an HR monitor (H7, Polar Electro Oy, Kempele, Finland). The integral of VO2 (L) and VCO2 (L) and the maximum 6-s moving average of relative VO2 (mL/kg.min), VE (L/min) and HR (bpm) were calculated for each set.

Muscle oxygenation: Throughout the protocol, oxygenated (O2Hb) and deoxygenated haemoglobin (HHb) were continuously monitored with a near-infrared spectroscopy device (Niro-200NX, Hamamatsu Phototonics, Hamamatsu, Japan) according with the manufacturer specifications. The integrals of O2Hb and HHb were calculated for each set of the protocol.

Neuromuscular fatigue assessment: Athletes executed a countermovement jump (CMJ) in a contact mat (Chronojump BoscoSystem, Software Version 2.2.0, Barcelona, Spain) before and after the exercise protocol, accessing values of jump height (JH). Three jumps were performed, separated by 30 s of rest, and the best jump was considered for analysis.

Data analysis: Power and sample calculations (G-Power, Version 3.1.9.2, Düsseldorf, Germany) were based on an effect size of 0.88 (McNaughton et al., 1997) for total work performed in the sprints, a power of 0.85 and a significance of 0.05. After the recruitment process, 12 athletes volunteered to participate in the study. One volunteer withdrew due to injury, leading to a sample size of 11 athletes. Statistical analysis was performed using the Statistical Package for the Social Sciences (IBM Corp, SPSS v27.0, Armonk, NY, USA) and R software (v4.2.0, Open-Source Code, General Public License). Normal distribution and sphericity were tested using Shapiro-Wilk's and Mauchly's tests, respectively. For variables with normal distribution, data was analysed using a two-way analysis of variance (ANOVA). Whenever a statistical significance was observed in the two-way ANOVA, post-hoc paired comparisons were performed with the Bonferroni correction. Statistical significance was set at p < 0.05. If normal distribution was not verified, the nparLD module of the R software was used to perform a non-parametric two-way ANOVA-type test and if any significant result was observed, a Friedman test and the post-hoc paired comparisons with the Bonferroni correction as well as a Wilcoxon test were performed. Statistical significance was adjusted according with the number of tests performed for each factor.

ELIGIBILITY:
Inclusion Criteria:

* Football players
* Regularly training with a weekly microcycle consisting of 3 to 5 training sessions and 1 game at the weekend
* Able to provide informed consent

Exclusion Criteria:

* Injury occurrence in the month previous to data collection
* Ergogenic supplements consumption in the month previous to data collection
* Having known intolerance to sodium bicarbonate

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Peak power output | 3 minutes through each set of the repeated sprints tasks
  Watt
Mean power output | 3 minutes through each set of the repeated sprints tasks
  Watt
Total Work | 3 minutes through each set of the repeated sprints tasks
  Joule
Sprint Decrement | 3 minutes through each set of the repeated sprints tasks
  percentage of power decrease

SECONDARY OUTCOMES:
Countermovement jump height | Before and after each repeated sprints tasks
  cm
Lactate accumulation | Before the repeated sprints tasks, between sets of the repeated sprints tasks, immediatly after the repeated sprints tasks, 2 minutes after the repeated sprints tasks
  mmol.L-1
Oxygen uptake | 3 minutes through each set of the repeated sprints tasks
  mL/kg.min
carbon dioxide production | 3 minutes through each set of the repeated sprints tasks
  Total L
Ventilation | 3 minutes through each set of the repeated sprints tasks
  L/min
Heart rate | 3 minutes through each set of the repeated sprints tasks
  bpm
Changes in muscle oxygenated haemoglobin | 3 minutes through each set of the repeated sprints tasks
  Absorvance relative to rest obtained by Near InfraRed Spectroscopy
Changes in muscle deoxygenated haemoglobin | 3 minutes through each set of the repeated sprints tasks
  Absorvance relative to rest obtained by Near InfraRed Spectroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Human Kinetics, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No